CLINICAL TRIAL: NCT06081257
Title: The Effect of "KB-120" Small Molecular Nutrient in Women With Decreased Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20230158-R
Record Dates: First submitted 2023-06-14; First posted 2023-10-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-06

CONDITIONS: Diminished Ovarian Reserve
MeSH Terms: interventions — Vitamin E

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): "KB-120" small molecule nutrients, taken orally once a day in one bag (30ml), and vitamin E100mg taken orally 2 times a day for a total of 3 menstrual cycles
  Interventions: Dietary Supplement: "KB-120" small molecular nutrient and vitamin E; Dietary Supplement: Vitamin E
- control group (Active Comparator): Vitamin E100mg is taken orally twice a day for a total of 3 menstrual cycles
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: "KB-120" small molecular nutrient and vitamin E — The experimental group was given oral "KB-120" small molecular nutrients, once a day, once a bag (30ml), and vitamin E100mg orally twice a day for a total of 3 menstrual cycles
  Arms: experimental group
Dietary Supplement: Vitamin E — Vitamin E100mg is taken orally twice a day for a total of 3 menstrual cycles

SUMMARY:
"KB-120" small molecular nutrient is a structural multi-molecular natural nutrient with different components. It is produced from strains and natural plant culture-medium that can be used in food and is designed according to different efficacy of different products by multi-stage solid-liquid complex fermentation technology. The functional directions of the product series involved are: immune function damage repair, intestinal villi damage repair, sperm development machinery damage repair, ovarian function damage repair, liver function damage repair, sleep disorder function damage repair, etc.Previous studies have shown that "KB-120" has good clinical effects on improving the number and function of male germ cells.Luanbao "KB-120" is a compound plant health drink specially for women. This study intends to give "KB-120" small molecule nutrients as nutritional supplement intervention in female patients with ovarian dysfunction, and observe its influence on endocrine function, ovarian reserve function and fertility in patients with ovarian dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with low ovarian function: FSH ≥10IU/L or AMH ≤1.1ng/ml.
2. The age at the time of signing the informed consent is 20-40 years old (including 20 and 40 years old) and has not been menopausal;
3. Be willing to sign written informed consent and comply with the study protocol

Exclusion Criteria:

1. Patients with severe anemia or malignant tumor; Lactation or pregnancy;
2. Eating disorders or anorexia;
3. Taking hormone drugs or participating in any other study.
4. There are factors that researchers believe cannot be included in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum FSH 1 | on the 3rd day of the 2nd menstruation（each cycle is 23-30 days）
  Blood samples were collected on the 3rd day of the 2nd menstruation
Concentration of serum FSH 2 | on the 3rd day of the 4th menstruation（each cycle is 23-30 days）
  Blood samples were collected on the 3rd day of the 4th menstruation
Concentration of serum AMH 1 | on the 3rd day of the 2nd menstruation（each cycle is 23-30 days）
  Blood samples were collected on the 3rd day of the 2nd menstruation
Concentration of serum AMH 2 | on the 3rd day of the 4th menstruation（each cycle is 23-30 days）
  Blood samples were collected on the 3rd day of the 4th menstruation

SECONDARY OUTCOMES:
The number of days of the menstrual cycle 1 | At the end of Cycle 1 （each cycle is 23-30 days）
  The number of days of the menstrual cycle 1
The number of days of the menstrual cycle 3 | At the end of Cycle 3（each cycle is 23-30 days）
  The number of days of the menstrual cycle 3
The diameter of dominant follicle and the number of days required for ovulation 1 | At the end of Cycle 1 （each cycle is 23-30 days）
  The follicle development of patients was monitored by ultrasound during the 1st menstrual cycle, and the monitoring interval was determined according to the clinical experience of clinicians and the development of patients' follicles
The diameter of dominant follicle and the number of days required for ovulation 2 | At the end of Cycle 3 （each cycle is 23-30 days）
  The follicle development of patients was monitored by ultrasound during the 3rd menstrual cycle, and the monitoring interval was determined according to the clinical experience of clinicians and the development of patients' follicles
pregnancy rate for women trying to get pregnant 1 | At the end of Cycle 1 （each cycle is 23-30 days）
  pregnancy rate for women trying to get pregnant
pregnancy rate for women trying to get pregnant 2 | At the end of Cycle 3 （each cycle is 23-30 days）
  pregnancy rate for women trying to get pregnant